CLINICAL TRIAL: NCT04719689
Title: Comparison of Dry Needling and Dry Cupping in Positional Fault of Pelvis Due to Myofascial Trigger Points in Quadratus Lumborum
Brief Title: Comparison of Dry Needling and Dry Cupping in Positional Fault of Pelvis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/20/0101 Huma Akhtar
Record Dates: First submitted 2021-01-10; First posted 2021-01-22 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Myofascial Trigger Point Pain; Quadratus Lumborum Syndrome; Positional Fault of Pelvis; Myofascial Trigger Point in Quadratus Lumborum
Keywords: Dry needling; Dry cupping; Quadratus lumborum
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling (Experimental): Dry needling, hot pack, stretching exercises.
  Interventions: Other: Dry needling
- Dry Cupping (Experimental): Dry cupping, hot pack, stretching exercises.
  Interventions: Other: Dry cupping

INTERVENTIONS:
Other: Dry needling — Experimental group 1 got this intervention containing Dry needling for 10 mins, followed by conventional physiotherapy treatment (hot pack and stretching) for 15 mins. Participants were treated 6 times over a 3 week period with 2 treatment sessions per week per patient. Pre and Post treatment readings were taken in 1st and 6th session over a 3 week period respectively. A follow up reading was also taken after 1 month for checking prolonged post treatment effects. Assessment was done via Pressure pain threshold Scale, Pelvic goniometer and Measuring tape for assessing functional positional fault of pelvis and muscle length of Quadratus lumborum
  Arms: Dry needling
Other: Dry cupping — Experimental group 2 got this intervention containing Dry cupping for 10 mins, followed by conventional physiotherapy treatment (hot pack and stretching) for 15 mins. Participants were treated 6 times over a 3 week period with 2 treatment sessions per week per patient. Pre and Post treatment readings were taken in 1st and 6th session over a 3 week period respectively. A follow up reading was also taken after 1 month for checking prolonged post treatment effects. Assessment was done via Pressure pain threshold Scale, Pelvic goniometer and Measuring tape for assessing functional positional fault of pelvis and muscle length of Quadratus Lumborum
  Arms: Dry Cupping

SUMMARY:
This project was a Randomized clinical trial conducted to Compare the effects of dry needling and dry cupping in Positional fault of pelvis due to Myofascial trigger points in Quadratus Lumborum so that we can have best treatment option for patients with myofascial trigger points.

DETAILED DESCRIPTION:
Non Probability Convenient sampling was done. Patients following eligibility criteria from Physiotherapy department of Islam Central hospital, Sialkot were considered. Sample size was calculated with Epitool calculator. 26 Participants were randomly allocated in two groups equally via convenient sampling method. Baseline assessment was done initially. Group A was given Dry needling technique and Group B was given Dry Cupping along with conventional physiotherapy treatment (hot pack and stretching). Duration of research was almost 6 months. Participants were treated 6 times over a 3 week period with 2 treatment sessions per week per patient. Pre and Post treatment readings were taken in 1st and 6th session over a 3 week period respectively. A follow up reading was also taken after 1 month for checking prolonged post treatment effects. Assessment was done via Pressure pain threshold Scale, Pelvic goniometer and Measuring tape for assessing functional positional fault of pelvis and muscle length of Quadratus Lumborum. All participants were provided written informed consent prior to commencement of the procedures. They were free to quit the treatment at any stage of research. Data was analyzed by using SPSS version 23.

ELIGIBILITY:
Inclusion Criteria:

* On palpation the presence of at least 1 active trigger point in quadratus lumborum. So the patient presents with low back pain.
* Patients presents with positional fault of pelvis (lateral tilt)(4).
* Patients having chronic Low Back Pain for at least more than 6 months(3).
* Patients agree to get treatment sessions for the research work.

Exclusion Criteria:

* Participants should not have taken any medications like analgesics, anti-coagulants, Non-steroidal anti-inflammatory drugs or muscle relaxants during this study or even 3 days before this study.
* Participants should not have received any other treatment for the pain management, because it will affect the results of the study.
* Patients with bleeding disorders, local or systemic infection, acute muscle trauma.
* Patients with comorbid conditions.
* Patients with severe physical disability and true leg length discrepancy(1).
* Pregnant females

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Change in Pain by 'Pressure Pain Algometer' | Baseline, 6th session(at 3rd week), follow up session after 1 month
  Change in Pain from baseline was checked at 6th session by Pressure Pain Algometer. A follow up reading was also taken after 1 month for checking prolonged post treatment effects.
Change in Range of Motion of lumbar spine side flexion by 'Goniometer' | Baseline, 6th session(at 3rd week), follow up session after 1 month
  Change in ROM from baseline was measured at 6th session. A follow up reading was taken after 1 month for checking prolonged post treatment effects. A goniometer is a device that measures an angle or permits rotation of an object to a definite position

SECONDARY OUTCOMES:
Change in pain by 'Numeric Pain Rating Scale' | Baseline, 6th session(at 3rd week), follow up session after 1 month
  Change in pain from baseline was measured at 6th session. A follow up reading was taken after 1 month for checking prolonged post treatment effects. The Numerical Pain Rating Scale (NPRS) is an 11 point pain scale that is completed by a patient himself, under the supervision of researcher.
Change in Range of Motion of lumbar side flexion by Measuring tape | Baseline, 6th session(at 3rd week), follow up session after 1 month
  Change in ROM from baseline was measured at 6th session. A follow up reading was taken after 1 month for checking prolonged post treatment effects. The method for using a tape measure to examine lateral flexion of the spine has been introduced in the literature.

CONTACTS AND LOCATIONS:
Overall Officials: Rabiya Noor, PhD, Principal Investigator — Riphah International University
Locations (1):
- Riphah IU, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pavkovich R. EFFECTIVENESS OF DRY NEEDLING, STRETCHING, AND STRENGTHENING TO REDUCE PAIN AND IMPROVE FUNCTION IN SUBJECTS WITH CHRONIC LATERAL HIP AND THIGH PAIN: A RETROSPECTIVE CASE SERIES. Int J Sports Phys Ther. 2015 Aug;10(4):540-51. PMID 26347305
- [Background] Kalichman L, Vulfsons S. Dry needling in the management of musculoskeletal pain. J Am Board Fam Med. 2010 Sep-Oct;23(5):640-6. doi: 10.3122/jabfm.2010.05.090296. PMID 20823359
- [Background] Haake M, Muller HH, Schade-Brittinger C, Basler HD, Schafer H, Maier C, Endres HG, Trampisch HJ, Molsberger A. German Acupuncture Trials (GERAC) for chronic low back pain: randomized, multicenter, blinded, parallel-group trial with 3 groups. Arch Intern Med. 2007 Sep 24;167(17):1892-8. doi: 10.1001/archinte.167.17.1892. PMID 17893311
- [Background] Leetun DT, Ireland ML, Willson JD, Ballantyne BT, Davis IM. Core stability measures as risk factors for lower extremity injury in athletes. Med Sci Sports Exerc. 2004 Jun;36(6):926-34. doi: 10.1249/01.mss.0000128145.75199.c3. PMID 15179160